CLINICAL TRIAL: NCT01762371
Title: Interdisciplinary Evaluation of Acute Effects From Khalifa's Therapy at Patients With Fully Ruptured Anterior Cruciate Ligament (ACL).
Brief Title: Khalifa Acute Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Sandner-Kiesling , MD, Univ.Prof.Dr., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KhalSbg1
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Totally Ruptured Anterior Cruciate Ligament in the Knee
Keywords: ACL; Knee; Ligament; Cruciate; Anterior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- K-Pat (Experimental): Getting one time one hour of Khalifa's therapy for ACL injury treatment.
  Interventions: Other: Khalifa Therapy

INTERVENTIONS:
Other: Khalifa Therapy — One hour of Khalifa's therapy which is specially applied pressure to the skin.

SUMMARY:
The primary hypothesis is that Khalifa's therapy has different acute effects in various organ systems i.e. proprioceptive, neuro-muscular, endogenous dopamine system, etc. These effects might indicate the pathway of the therapy.

DETAILED DESCRIPTION:
According to our previous study that evaluated the efficacy of Khalifa's therapy the investigators have seen that the therapy has acute effects which resulted in better knee function and later even in better healing of the ACL injury. This study should clear exactly which effects and pathways are involved in the therapy from multiple (interdisciplinary) point of views. Therefore the investigators will measure parameters that might be associated with this special technique directly before and after the therapy.

ELIGIBILITY:
Inclusion Criteria:

* totally ruptured ACL - MRI verified, 2 weeks old as a maximum
* knee function: Any functional inhibition (stretching, bending or load)
* BMI: 18-25
* athletically active

Exclusion Criteria:

* any surgical procedures at the injured knee at any previous time
* any acute surgical indication
* diabetes mellitus and/or high blood pressure
* any permanent drug treatment

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Laser Doppler-Flow | 1 hour
  Perfusion
NIRS | 1 hour
  Near infrared spectroscopy, Oxygen saturation
IR Thermography | 1 hour
  Infrared thermography, temperature
QST | 1 hour
  Quantitative sensoric testing, pain
HRV | 1 hour
  Heart rate variability, sympathicus/parasympathicus activation
EEG | 1 hour
  Electroencephalogram, brain waves
Knee function | 1 hour
  IKDC Score KT-1000 test Clinical / physical examination
SportsScience | 2 hours
  Posturomed Motion capture proprioception muscle power range of motion
Blood | 1 hour
  Catecholamines endorphins standard blood parameters

SECONDARY OUTCOMES:
Questionnaire | 1 hour
  Different questions about pain, lifestyle, subjective parameters

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kastner, MD, Principal Investigator — AKH Linz; Andreas Sandner, MD, Principal Investigator — Med Uni Graz
Locations (1):
- Sports Center of University Salzburg, Hallein, Salzburg, Austria